CLINICAL TRIAL: NCT05971654
Title: Effect Of Azithromycin On Pregnancy Prolongation In Women at Risk of Preterm Labour
Brief Title: Effect Of Azithromycin in Women at Risk of Preterm Labour
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Azithromycin preterm
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Preterm Labor
Keywords: preterm delivery; Azithromycin
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Experimental): azithromycin.:500 mg PO once for 5 days every month
  Interventions: Drug: azithromycin
- control (No Intervention): pregnant woman at risk of preterm delivery

INTERVENTIONS:
Drug: azithromycin — azithromycin.:500 mg PO once for 5 days every month
  Other Names: zisrocin
  Arms: Azithromycin

SUMMARY:
The aim of this study is to evaluate the benefit of the addition of azithromycin to standard treatments to prolong pregnancy in women having intact membranes and is at risk of or in preterm labour.

DETAILED DESCRIPTION:
Study Design:

Comparative controlled study.

Study site :

The study will be conducted at the department of Obstetrics and Gynecology at Beni-Suef University Hospital.

Study period:

The study will be conducted from 15th September 2022 till reaching the target number.

Study Population The control group will include pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy.

The test group will involve pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy plus prophylactic azithromycin.:500 mg PO once for 5 days every month.

Sample size:

The sample size was determined using G*Power Version 3.1.9.2 [computer software] (Franz Faul, Kiel, Germany),Power analysis for a chi-square test was conducted in G-POWER to determine a sufficient sample size using an alpha error of probability of 0.05, power of 0.95, a medium effect size (w = 0.3) and 1 degree of freedom. Based on the aforementioned assumptions, the desired sample size is 145. By calculating 25% drop out, so the least total sample size in both groups will be 200 patients (95 patients in each group).

Each patient will be subjected to:

Thorough history taking and examination. Investigations: Complete blood picture (CBC), bleeding profile , kidney function tests and liver function tests will be done.

Ultrasound: 2D Ultrasound assessing :

It will be carried out in Gynecology and Obstetrics department in Beni-Suef University Hospital, ultrasonography criteria: Ultrasound biometry of the fetus is now the gold standard for assessing fetal growth. The measurements most commonly used are the biparietal diameter, head circumference, abdominal circumference and femur length

ELIGIBILITY:
Inclusion Criteria:

* 24 < Pregnancy <37 weeks of gestation.
* Threat or history of preterm labour.
* Preterm labour itself (Non established)

Exclusion Criteria:

* antibiotics use within 14 days (except for pericerclage prophylaxis, or streptococcus B prophylaxis);
* PPROM; and fetal extraction required <37 weeks.
* Current or past history of medical diseases (Diabetes Milletus, Hypertension, Systemic Lupus Erythematosus, Cardiac diseases, etc ).
* Adverse perinatal outcome due to abdominal trauma.
* Structural fetal anomalies detected during anomaly scan.
* Allergy to Azithromycin.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Gestational age at time of delivery | 9 months
  measured in week's days'number

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided